CLINICAL TRIAL: NCT02533934
Title: A Retrospective/Prospective Cohort Study to Assess Safety, Tolerability, and Efficacy of Sofosbuvir Based Direct Acting Antiviral (DAA) Therapy for Hepatitis C Treatment in HIV/HCV Coinfected Subjects Pre or Post Liver Transplant
Brief Title: Sofosbuvir Based DAA Therapy in HIV/HCV Coinfected Pre or Post Liver Transplant
Acronym: STOP-CO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Icahn School of Medicine at Mount Sinai (Other); Columbia University (Other); University of Pennsylvania (Other); University of Maryland, College Park (Other); Georgetown University (Other); Johns Hopkins University (Other); National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12044; 1U01AI115714 (NIH)
Record Dates: First submitted 2015-08-25; First posted 2015-08-27 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: HIV; Hepatitis C; Cirrhosis
Keywords: HIV; Hepatitis C; Liver Disease; HCV Treatment; transplant
MeSH Terms: conditions — Hepatitis C; Fibrosis; Liver Diseases | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Sofosbuvir based HCV Therapy (Experimental): Prospective and retrospective treatment for HCV
  Interventions: Drug: Harvoni

INTERVENTIONS:
Drug: Harvoni — Treatment of Hepatitis C with sofosbuvir based HCC therapy
  Other Names: SOF/LDV

SUMMARY:
Retrospective/Prospective, open-label study using sofosbuvir based DAA therapy to treat HIV/HCV coinfected pre or post liver transplant participants

DETAILED DESCRIPTION:
Approximately fifty HIV/HCV coinfected patients with decompensated liver disease will be enrolled in the study. Ten (up to twenty) subjects will be treated with FDC SOF/LDV pre or post liver transplant and followed prospectively. Forty + subjects will be enrolled retrospectively with the intent to capture all patients who have been exposed to sofosbuvir based DAA therapies at participating sites since 1/2014, and to mirror the population being enrolled prospectively.

In addition, participants in the retrospective arm will be contacted to consent to one prospective study visit for liver staging to determine rates of reversal of decompensation, reversal of cirrhosis and improvements in graft survival post treatment, and for future contact by the NIH Clinical Center to assess longer term outcomes when this study ends.

ELIGIBILITY:
RETROSPECTIVE ARM INCLUSION CRITERIA

The intent of the Retrospective Arm is to capture all HIV/HCV coinfected patients exposed to sofosbuvir based DAA therapy since 2014, to mirror the population enrolled in the Prospective Arm.

Liver transplant candidates (listed) and decompensated cirrhotics (not listed) for liver transplant

1. Treated with sofosbuvir based DAA for any duration since 2014
2. Age >18 years at time of treatment
3. Pre-treatment Child's Pugh score of 7 or greater
4. Pre-treatment laboratory MELD >=6 and <=0
5. Survived at least 12 weeks after start of treatment
6. HIV-positive on stable ART for at least 4 weeks pre-treatment
7. Chronic HCV infection with at least one measurement of plasma HCV RNA >= 1,000 IU/mL prior to treatment with sofosbuvir based DAA therapy
8. HCV genotype 1, 4, 5 or 6

Liver transplant recipients

1. Treated with sofosbuvir based DAA post liver transplant for any duration since 2014
2. Liver transplant from 2000 to current
3. Age >18 years at time of treatment
4. Treated initiated at least 1 month post-liver transplant
5. Post-LT stage of liver disease documented within the prior year of treatment start date by standard of care methods of liver staging
6. Survived at least 12 weeks after start of treatment
7. HIV-positive on stable ART for at least 4 weeks pre-treatment
8. Chronic HCV infection with at least one measurement of plasma HCV RNA >= 1,000 IU/mL prior to treatment with sofosbuvir based DAA therapy
9. Fibrosis staging done within 1 year of start of DAA therapy
10. HCV genotype 1, 4, 5 or 6

PROSPECTIVE ARM INCLUSION/EXCLUSION CRITERIA

Pre-liver transplant candidates

* Enrollment will be targeted to occur at least 12 weeks prior to anticipated transplant date.
* Screening laboratory MELD >=6 and <=20 (NIH) or <=30 (non-NIH sites)

Post-liver transplant recipients

* Recipients with evidence of recurrent HCV viremia
* Subjects with compensated and decompensated liver disease
* Screening laboratory MELD >=6 and <=20 (NIH) or <=30 (non-NIH sites)
* Life expectation of >12 weeks

Inclusion Criteria

1. Over 18 years of age at screening
2. Female participants of child bearing potential must have a negative urine pregnancy test at day 0 prior to dosing.
3. Has received a liver transplant for HCV or has decompensated cirrhosis (Child's Pugh score of 7 or greater)
4. Have HIV-1 infection and either:

   1. On HIV medications (antiretrovirals) for at least 4 weeks WITH

      * An HIV viral load less than the level of detection OR
   2. On no HIV medications for at least 8 weeks WITH:

      * A CD4 count of 500 cells/mm3 or more OR
      * HIV viral load of < 500 copies/mL with a stable CD4 count for at least 3 months
5. Chronic HCV infection as documented by at least one measurement of plasma HCV RNA >= 1,000 IU/mL during screening and at least one of the following:

   A positive anti-HCV antibody, HCV RNA, or an HCV genotype test at least 12 months prior to baseline (Day 0) visit together with positive HCV RNA test
6. HCV genotype 1, 4, 5 or 6
7. The use of an anti-HCV positive donor is allowed for participants who have detectable HCV RNA at the time of transplant.
8. The use of an HIV+ donor is allowed if the participant is enrolled in an IRB approved HOPE Act protocol at the transplant site. If the HIV+ donor is also HCV co-infected, then the recipient must have detectable HCV RNA at the time of transplant.
9. Able to effectively communicate with the Investigator and other center personnel.
10. Willing to give written informed consent and comply with the study restrictions and requirements.
11. Willingness to allow stored blood or tissue samples to be used in the future for studying liver disease and immune function.
12. Willingness to permit HLA typing to be performed.
13. Have a transplant team available for all primary and transplant-related care.
14. If not yet transplanted: expected to be at least 12 weeks prior to transplant in order to complete treatment course.
15. If not yet transplanted: Must have prior standard of care liver staging consistent with F4.
16. If not yet transplanted: For pre-LT patients with HCC, they must meet Milan criteria at time of enrollment to be eligible
17. If post-liver transplant, must be at least 1 month since transplant procedure to begin treatment.
18. If post-liver transplant, liver disease staging must be documented within the prior year by standard of care methods of liver staging

Exclusion Criteria

1. Positive HBsAg at screening.
2. History of any other clinically active chronic liver disease (e.g., hemochromatosis, autoimmune hepatitis, Wilson's disease, >=1 antitrypsin deficiency, alcoholic liver disease, and toxin exposures).
3. Treatment with unlicensed herbal/natural remedies suggested to be taken for hepatitis treatment, such as Milk thistle, St. Johns Wort or Cats Claw, within 28 days of start of treatment
4. Treatment with IFN, RBV, telaprevir or boceprevir or any other approved or experimental medication with known anti-HCV activity within 1 month prior to screening date
5. Any prior exposure to an HCV NS5a specific inhibitor
6. A personal history of or first degree relative with a history of Torsade de pointes.
7. Abnormal hematological and biochemical parameters, including:

   1. Hemoglobin < 8g/dL
   2. Estimated GFR, calculated by the CKD-EPI equation, <30 mL/min/ per 1.73 m2
   3. Sodium <120 mmol/L
8. History of major organ transplantation other than liver or kidney transplantation.
9. Difficulty with blood collection/poor venous access for phlebotomy that would prevent the collection of study required samples
10. Infection requiring systemic antibiotics at the time of screening
11. Active or recent history (≤ 6 months) of drug or alcohol abuse
12. Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug.
13. Donation or loss of more than 400 mL blood within 8 weeks prior to first dose administration.
14. Any medications prohibited (see table 2 in section 8.11) within 28 days prior to Day 0 visit and likely required during study treatment period
15. History of clinically significant drug allergy to nucleoside/nucleotide analogs.
16. History or current evidence of psychiatric illness, endocrine, immunologic disorder, pulmonary, cardiac disease, seizure disorder, cancer or other conditions that in the opinion of the investigator makes the patient unsuitable for the study. Chronic medical conditions, especially if treated with medications (such as hypertension), must be stable at the time of screening. No new therapies should be started within 28 days prior to the study that may confound the assessment of study drug safety.
17. Participation in a clinical study (other than an IRB approved HOPE Act protocol involving the utilization of an HIV+ donor) in which an investigational drug, biologic, or device was received within 12 weeks prior to first dose administration.
18. Pregnant/Breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stock, MD, PhD, Principal Investigator — University of California, San Francisco; Henry Masur, MD, Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: STOP-CO is a multi-center prospective and retrospective, open-label study using sofosbuvir-based DAA therapy to treat HIV/HCV coinfected participants pre- or post-LT.
Pre-assignment Details: The study was designed to prospectively assign ledipasvir-sofosbuvir to participants awaiting transplant or ≥1 month post-transplant. During the course of the trials, DAAs became widely available and the standard of care for the target study population. Only 7 participants could be enrolled in the prospective arm of this study with ledipasvir-sofosbuvir. Therefore in 2017 the study was amended to include retrospective participants treated with any sofosbuvir-based therapy after 2014.
Groups:
- Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant; Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant: The study was implemented at 7 designated sites across the United States. Participants were HIV-positive on a stable antiretroviral (ART) regimen for at least 4 weeks pre-treatment. The retrospective portion of the study enrolled participants treated with sofosbuvir-based DAAs for any duration since 2014 were eligible. HCV genotypes 1, 4, 5 or 6 were included with at least one serum HCV RNA ≥ 1000 IU/mL prior to treatment. Pre-LT participants had a pre-treatment Child's Pugh Turcotte (CPT) score ≥ 7 and a pre-treatment laboratory MELD ≥ 6 and ≤ 30 and included both listed LT candidates and participants who had decompensated cirrhosis not listed for LT. Inclusion criteria for post-LT participants were a LT after 2000 and DAA treatment initiated ≥ 1 month after LT. Prospective participants were accrued from 12/2016-11/2018. Additional exclusion criteria for prospective participants were chronic hepatitis B infection, a history of any other clinically active chronic liver disease, and prior treatment for HCV within one month of screening. Retrospective participants were enrolled between 4/2018 and 6/2019. Information about type of SOF-based therapy in the retrospective participants was not collected for this study.
Period: Overall Study
Arm/Group | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant | Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant
Started | 42 | 26
Completed | 42 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant | Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant | Total
Number analyzed (Participants) | 42 | 26 | 68
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 56.4 [52.7 to 60.4] | 57.2 [52.6 to 61.7] | 56.6 [52.3 to 61.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 31 | 22 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 11 | 32
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 42 | 26 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR)
Description: Sustained virologic response (SVR) defined by hepatitis C virus (HCV) RNA less than the lower level limit of quantification (LLOQ) of <15 IU/ml at a median time of 38.5 months after the end of sofosbuvir-based direct-acting antiviral (DAA) therapy
Time Frame: Median time from end of treatment was 38.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant | Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant
Number analyzed (Participants) | 42 | 26
Participants | 38 | 25

2. Secondary Outcome: Reversal in Decompensation
Description: Number of participants with an improved, worsened or unchanged MELD (Model for End-stage Liver Disease) score. A MELD score ranges from 6 to 40. The higher the number, the worse the liver disease.
Time Frame: Median months from baseline to last MELD measurement is 48 months
Population: participants treated pre-liver transplant, who had MELD scores available pre and post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant
Number analyzed (Participants) | 33
Participants
  Participants who MELD score improved from baseline | 19
  Participants who MELD score worsened from baseline | 11
  Participants who MELD score was unchanged | 3

3. Secondary Outcome: Change in Liver Fibrosis
Description: Change in AST to Platelet Ratio Index (APRI) where negative values indicate improvement in liver fibrosis score and positive values indicate worsening of fibrosis score. There is no upper or lower limit for change.
  Change in Fibrosis-4 (FIB-4) where negative values indicate improvement in liver fibrosis score and positive values indicate worsening of fibrosis score. There is no upper or lower limit for change.
Time Frame: Median months from baseline to last APRI measurement is 41 months Median months from baseline to last FIB-4 measurement is 41 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant | Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant
Number analyzed (Participants) | 42 | 26
units on a scale
  Change in AST to platelet ratio index (APRI) | -0.71 [-1.63 to -0.37] | -0.72 [-1.41 to -0.39]
  Change in Fibrosis-4 (FIB-4) | -2.76 [-4.78 to -0.47] | -1.06 [-2.04 to -0.20]
Statistical Analysis 1: Comparison: Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant; APRI change from baseline to last follow-up; Test type: Equivalence — Equivalence margin is defined by the a priori threshold for statistical significance; p < .01, Kruskal-Wallis
Statistical Analysis 2: Comparison: Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant; APRI change from baseline to last follow-up; Test type: Equivalence — Equivalence margin is defined by the a priori threshold for statistical significance; p < .01, Kruskal-Wallis
Statistical Analysis 3: Comparison: Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant; FIB4 change from baseline to last follow-up; Test type: Equivalence — Equivalence margin is defined by the a priori threshold for statistical significance; p < .01, Kruskal-Wallis
Statistical Analysis 4: Comparison: Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant; FIB4 change from baseline to last follow-up; Test type: Equivalence — Equivalence margin is defined by the a priori threshold for statistical significance; p < .01, Kruskal-Wallis

4. Secondary Outcome: HIV Viral Breakthrough or Relapse
Description: Number of participants with a detectable HIV viral load after sofosbuvir-based HCV therapy
Time Frame: Median months from baseline to last HIV follow-up is 38 months
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant | Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant
Number analyzed (Participants) | 42 | 26
Participants | 0 | 0

5. Secondary Outcome: Number of Subjects Treated With Sofosbuvir-based DAA Therapy Who Had Alanine Aminotransferase (ALT) Normalization Post Treatment (Normal Reference Range: 7 - 55 IU/L)
Description: Change in ALT after sofosbuvir based DAA therapy
Time Frame: Median months from baseline to last ALT measurement is 41 months
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant | Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant
Number analyzed (Participants) | 40 | 26
Participants | 31 | 20
Statistical Analysis 1: Comparison: Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant; Test type: Equivalence — Equivalence margin is defined by the a priori threshold for statistical significance; p < 0.001, Wilcoxon (Signed Rank Test)

ADVERSE EVENTS:
Time Frame: Prospective Subjects: from participants first dose until 6 months post treatment discontinuation, through study completion, up to twelve months, plus deaths at any-time. Retrospective Subjects: from participants first dose to end of treatment, through study completion, up to six months, plus deaths at any-time.
Description: All serious adverse events were recorded from time of HCV treatment initiation until last followup for subjects enrolled prospectively (7). For subjects enrolled retrospectively (61), only serious adverse events related to hospitalizations during treatment with sofosbuvir based DAA therapy, anemia require transfusion or EPO during treatment with DAA therapy, or death were recorded.
Arm/Group | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant | Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant
All-Cause Mortality (participants affected / at risk) | 10/42 | 3/26
Serious Adverse Events (participants affected / at risk) | 18/42 | 7/26
Other Adverse Events (participants affected / at risk) | 2/42 | 4/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant (N=42) | Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant (N=26)
Hospitalization (Unknown) (General disorders) | 3 (5) | 0 (0) — Reported hospitalization with unknown etiology in retrospective study participant
Hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) — abnormal movements, hyperactivity, etiology unknown
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) — infection AKI
Ampullary stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
DVT (Vascular disorders) | 0 (0) | 1 (1) — Deep vein thrombosis
Dyspnea (Vascular disorders) | 1 (1) | 0 (0)
esophagogastroduodendoscopy (Hepatobiliary disorders) | 2 (2) | 0 (0) — due to cirrosis
Gasteroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gout (Immune system disorders) | 1 (1) | 0 (0)
Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) — scheduled hospitalization for followup surgery to remove polyps from colon
Hyperglycemic seizure (Hepatobiliary disorders) | 1 (1) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Neck femur fracture (General disorders) | 1 (1) | 0 (0)
Polysubstance use (Psychiatric disorders) | 1 (1) | 0 (0)
Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — right upper extremity clot
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive with hypoactive delirium (Nervous system disorders) | 0 (0) | 1 (1)
Ventral hernia (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults With HIV and Chronic HCV and End-stage Liver Disease (ESLD) Pre-liver Transplant (N=42) | Adults With HIV With Chronic HCV and Any Stage of Liver Disease Post-liver Transplant (N=26)
Nausea (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Vomiting (General disorders) | 0 (0) | 1 (1)
Headaches (General disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperbilirubiinemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pnemonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was limited by the necessity to change the design from a prospective to a retrospective/prospective analysis. This change in study design resulted from the urgency in treating the HIV/HCV coinfected liver transplant candidate with DAAs, based on the dismal survival outcome in this cohort. By the time this trial was approved, many of the DAAs for HCV were approved, and centers immediately treated their decompensated HIV/HCV recipients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02533934/Prot_SAP_000.pdf
  • Informed Consent Form: Retrospective Informed Consenst (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02533934/ICF_001.pdf
  • Informed Consent Form: Prospective Informed Consent (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02533934/ICF_002.pdf